CLINICAL TRIAL: NCT01276171
Title: Ultrasound-image Guided Versus Doppler Guided Versus Palpation Technique for Arterial Cannulation in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Kenichi Ueda, Clinical Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201001776
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-04

CONDITIONS: Anesthesia
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ultrasound (Active Comparator): Participants will place arterial line using ultrasound technique
  Interventions: Procedure: Ultrasound
- Doppler (Active Comparator): Participants will place arterial line using doppler technique
  Interventions: Procedure: Doppler
- Palpation (Active Comparator): Participants will place arterial line using palpation technique
  Interventions: Procedure: Palpation

INTERVENTIONS:
Procedure: Ultrasound — Participants will place arterial line using ultrasound technique
  Arms: Ultrasound
Procedure: Doppler — Participants will place arterial line using doppler technique
  Arms: Doppler
Procedure: Palpation — Participants will place arterial line using Palpation technique
  Arms: Palpation

SUMMARY:
Radial arterial cannulation is a common invasive procedure for real-time measurement of arterial blood pressure. Placement of the arterial catheter using conventional palpation is often relatively easy and quick, but this is not always true. A relatively new method for direct visualization of the artery is the use of two-dimensional ultrasound. This technique allows cannulation of the artery to take place under real-time visualization and may increase the success rate of first time pass of the needle. Another technique utilizing Doppler has also proven to be effective in cannulating the radial artery. This technique utilizes changes in acoustic pitch as the probe passes directly over the artery. The primary objective of this study is to compare the first attempt success rate for radial artery cannulation among the palpation, Doppler and U/S guided technique when applied by trainees. Secondary outcomes include: success rate within 5 minutes, successful, number of attempts required, and correlation between success rate and operator experience for successful cannulation of the radial artery.

DETAILED DESCRIPTION:
Radial artery cannulation is a common invasive procedure in the operating room, intensive care unit and emergency department. It allows continuous hemodynamic monitoring and repeated arterial blood sampling. Although severe complications are rare, successful radial artery cannulation can be technically challenging, particularly in hypotensive patients and those with vascular disease. Multiple unsuccessful attempts at arterial cannulation increase patient discomfort, delay timely care and may also contribute to adverse events such as arterial spasm or local hematoma.

The radial artery is traditionally located by palpation. A number of techniques to aid radial artery localization have been described. Doppler-assisted radial arterial cannulation was first described in 1976. Several case reports suggest that Doppler can be helpful in patients with difficult arterial access. More recently, ultrasound-guided radial artery cannulation has been described. In a recent meta-analysis of four randomized controlled trials, ultrasound increased the rate of cannulation on the first attempt by 71% compared with palpation. However, two of the studies were of children and all four were small, with 30-152 participants (311 in total), making the generalizability of these results to adult patients uncertain. Furthermore, variation in the training and experience of the operators was evident within one of the studies.

Accordingly, the aim of this study is to compare three different radial arterial cannulation techniques in adult surgical patients when performed by anesthesia residents: Doppler; palpation; and ultrasound. We think that ultrasound would have a higher rate of cannulation on the first attempt compared with other techniques.

ELIGIBILITY:
Inclusion Criteria:

* Main OR patients at UIHC who require arterial catheter placement for surgery

Exclusion Criteria:

* The patients who will be excluded from the study include those who have had arterial cannulation in the previous month, infections at site of insertion, and AV shunts in upper extremity.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 749 (Actual)
Dates: Start 2010-02; Primary Completion 2011-12 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Ueda, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
We are not planning on sharing IPD.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound | Doppler | Palpation
Started | 249 | 244 | 256
Completed | 249 | 244 | 256
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound | Doppler | Palpation | Total
Number analyzed (Participants) | 249 | 244 | 256 | 749
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 148 | 144 | 157 | 449
  >=65 years | 101 | 100 | 99 | 300
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [48 to 71] | 61 [51 to 72] | 59 [50 to 70] | 60 [50 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 107 | 106 | 319
  Male | 143 | 137 | 150 | 430
Region of Enrollment [Number; unit: participants]
  United States | 249 | 244 | 256 | 749

OUTCOME MEASURES:

1. Primary Outcome: First Attempt Success Rate With 3 Different Technique
Description: The primary objective of this study is to compare the first attempt success rate for radial artery cannulation between the palpation, Doppler and U/S guided technique when applied by anesthesia trainees. Secondary outcomes include: success rate within 5 minutes, time to successful cannulation compared with three different techniques.
Time Frame: 5 minutes
Measure: Number; unit: participants
Arm/Group | Ultrasound | Doppler | Palpation
Number analyzed (Participants) | 249 | 244 | 256
participants | 132 | 101 | 96

2. Secondary Outcome: Time to Successful Cannulation
Time Frame: 5 minutes
Measure: Median (Inter-Quartile Range); unit: min
Arm/Group | Ultrasound | Doppler | Palpation
Number analyzed (Participants) | 249 | 244 | 256
min | 32 [19 to 51] | 118 [69 to 198] | 91 [60 to 153]

3. Secondary Outcome: Total Success Rate
Time Frame: 5 min
Population: chi-squre test
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrasound | Doppler | Palpation
Number analyzed (Participants) | 249 | 244 | 256
Participants | 170 | 147 | 160

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Ultrasound | Doppler | Palpation
Serious Adverse Events (participants affected / at risk) | 0/249 | 0/244 | 0/256
Other Adverse Events (participants affected / at risk) | 27/249 | 22/244 | 29/256
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrasound (N=249) | Doppler (N=244) | Palpation (N=256)
Hematoma (Blood and lymphatic system disorders) | 27 (27) | 22 (22) | 29 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes